CLINICAL TRIAL: NCT03528538
Title: The Efficacy of Fenugreek Supplementation on Men's Health: A Randomized Controlled Trial
Brief Title: The Efficacy of Fenugreek Supplementation on Men's Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacksonville University (Other)
Collaborators: SPECNOVA LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JUFenugreek2018
Record Dates: First submitted 2018-02-26; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Aging; Testosterone Deficiency
Keywords: Fenugreek; Aging Male Symptoms; Testosterone; Supplementation; Double Blind; Body Composition

STUDY DESIGN:
Intervention Model Description: Subjects will complete 3 assessments during the study at Day 0, Week 4, and Week 8. At each assessment, they complete the following: self-report inventories (e.g., Aging Male Symptoms Questionnaire, Trait Anxiety Inventory, Health-related Quality of Life), body composition via BOD POD, heart rate, blood pressure, and blood draws. The subjects will be randomized to one of the following three conditions: (1) AlphaFenTM fenugreek (400 mg/d), (2) AlphaFenTM fenugreek (500 mg/d), or (2) placebo control. The subjects will be asked to take one capsule of the fenugreek supplement or placebo daily for eight weeks.
Who Masked: Participant, Investigator
Masking Description: The investigators and the participants remained blind until after the total completion of the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- AlphaFen fenugreek 400 mg (Active Comparator): This group received 400 mg of fenugreek to be ingested daily for 60 days.
  Interventions: Dietary Supplement: AlphaFen fenugreek 400 mg
- AlphaFen fenugreek 500 mg (Active Comparator): This group received 500 mg of fenugreek to be ingested daily.
  Interventions: Dietary Supplement: AlphaFen fenugreek 500 mg

INTERVENTIONS:
Dietary Supplement: AlphaFen fenugreek 400 mg — A brand of fenugreek supplementation that was produced by SPECNOVA. Pure fenugreek without any additives.
  Arms: AlphaFen fenugreek 400 mg
Dietary Supplement: AlphaFen fenugreek 500 mg — A brand of fenugreek supplementation that was produced by SPECNOVA. Pure fenugreek without any additives.
  Arms: AlphaFen fenugreek 500 mg
Other: Placebo — rice flour in a vegetable/ cellulose capsule
  Arms: Placebo

SUMMARY:
1. The problem: There is limited research on the use of herbal supplements in general, and fenugreek specifically, to improve male health, particularly to increase testosterone levels. As well, no located studies have examined the effects of fenugreek supplementation on healthy men's health-related quality of life, anxiety levels, and body composition.
2. Relevant research examined the effects of fenugreek supplementation with healthy men aged between 43 and 70 years of age. The researchers found that both total serum testosterone and free testosterone increased compared to placebo after 12 weeks of active treatment. The researchers concluded that fenugreek supplementation was a safe and effective treatment for reducing symptoms of possible androgen deficiency, improves sexual function and increases serum testosterone in healthy middle-aged to older men. Another study found that fenugreek supplementation improved aging male symptoms and testosterone levels remained in a normal range in healthy men aged 25 to 45 years.
3. The importance of this study: The importance of this study is to help determine if fenugreek supplementation affects testosterone levels, body composition, health-related quality of life, anxiety, and aging symptoms in healthy men aged 21 - 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men between the ages of 21- 45 that were recreationally active.

Exclusion Criteria:

* Above 30% body composition, not in the age range, history of asthma, diabetes, hypoglycemia, or took any hormonal supplements such as testosterone or anabolic steroids.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life Questionnaire | 8 weeks
  The Centers for Disease Control (CDC) Health-related Quality of Life measure will be used to assess health-related quality of life. This scale has excellent psychometric properties. The HRQoL assesses the positive and negative aspects of a person's life such as satisfaction or distress and the impact of these factors to their perceived health and life experience. This questionnaire is a valid and reliable measure than can be used to evaluate the individuals physical and mental perceptions.
Aging Male Symptoms Questionnaire | 8 weeks
  The Aging Male Questionnaire consists of 17 questions in 3 sub-scales (i.e., psychological, somatic and sexual) that assesses symptoms of aging specific for men. These sub-scales as well as the total score were used to assess symptoms. Having symptoms from the AMS questionnaire merely suggests a male may have deficiencies but blood samples are the best determinants of this condition. The higher the score, the worst the outcome.
Blood | 8 weeks
  From 10 mL of fasted blood. The free testosterone, total testosterone, and estradiol levels will be extracted from the blood sample.
Body Composition | 8 weeks
  The BODPOD machine is considered the gold standard for body composition as it has a range of error between ± 1 to 2.7% and is easier to complete than underwater weighing. The BODPOD was used to observe body composition at each assessment
Strength | 9 weeks
  Hand grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hausenblaus, PhD, Principal Investigator — Jacksonville University
Locations (1):
- Jacksonville University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daig I, Heinemann LA, Kim S, Leungwattanakij S, Badia X, Myon E, Moore C, Saad F, Potthoff P, Thai do M. The Aging Males' Symptoms (AMS) scale: review of its methodological characteristics. Health Qual Life Outcomes. 2003 Dec 15;1:77. doi: 10.1186/1477-7525-1-77. PMID 14675485
- [Background] Dempster P, Aitkens S. A new air displacement method for the determination of human body composition. Med Sci Sports Exerc. 1995 Dec;27(12):1692-7. PMID 8614327
- [Background] Fess, E. E. (1992). Grip strength. In clinical assessment recommendations. 2nd ed. Chicago: American Society of Hand Therapists.
- [Background] Rao A, Steels E, Inder WJ, Abraham S, Vitetta L. Testofen, a specialised Trigonella foenum-graecum seed extract reduces age-related symptoms of androgen decrease, increases testosterone levels and improves sexual function in healthy aging males in a double-blind randomised clinical study. Aging Male. 2016 Jun;19(2):134-42. doi: 10.3109/13685538.2015.1135323. Epub 2016 Jan 20. PMID 26791805
- [Background] Spielberger, CD., Gorsuch, R.L., Lushene, R., Vagg, P.R., & Jacobs, G.A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Steels E, Rao A, Vitetta L. Physiological aspects of male libido enhanced by standardized Trigonella foenum-graecum extract and mineral formulation. Phytother Res. 2011 Sep;25(9):1294-300. doi: 10.1002/ptr.3360. Epub 2011 Feb 10. PMID 21312304
- [Background] Wankhede S, Mohan V, Thakurdesai P. Beneficial effects of fenugreek glycoside supplementation in male subjects during resistance training: A randomized controlled pilot study. J Sport Health Sci. 2016 Jun;5(2):176-182. doi: 10.1016/j.jshs.2014.09.005. Epub 2015 Mar 7. PMID 30356905
- [Background] Zack MM; Centers for Disease Control and Prevention (CDC). Health-related quality of life - United States, 2006 and 2010. MMWR Suppl. 2013 Nov 22;62(3):105-11. PMID 24264499
- [Derived] Hausenblas HA, Conway KL, Coyle KRM, Barton E, Smith LD, Esposito M, Harvey C, Oakes D, Hooper DR. Efficacy of fenugreek seed extract on men's psychological and physical health: a randomized placebo-controlled double-blind clinical trial. J Complement Integr Med. 2020 May 22;18(2):445-448. doi: 10.1515/jcim-2019-0101. PMID 32441668